CLINICAL TRIAL: NCT02016651
Title: Positioning and Gastric Aspiration in Ventilated Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Aly, Visiting Professor of Pediatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20120101
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Respiratory Aspiration of Gastric Contents
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right side position (Experimental): Premature infants on mechanical ventilation are kept on their right side
  Interventions: Behavioral: Right side position
- Supine position (No Intervention): Premature infants on mechanical ventilation are kept on their back

INTERVENTIONS:
Behavioral: Right side position — Enrolled infants are positioned on their back or right side. Tracheal aspirate is assessed for pepsin concentration as an index of aspiration.
  Arms: Right side position

SUMMARY:
Gastro-esophageal reflux and aspiration is a common problem in premature infants receiving mechanical ventilation. Pepsin measured in tracheal aspirate (TA) emerged as a specific marker for aspiration. The objective of this study is to examine if TA pepsin will change when ventilated premature infants are positioned in two different positions; on their back vs. on their right side.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 28 and 32 weeks gestational age
* postnatal age > 72 hours
* tracheally intubated and receiving conventional mechanical ventilation
* feeding enterally more than 20 ml per day.

Exclusion Criteria:

* neurological insult in the form of perinatal asphyxia (pH <7, base deficit more than 12, Apgar score at < 3 at 5 minutes of life), intracranial hemorrhage grades 3 or 4 at 72 hours of age or periventricular leucomalacia
* major congenital anomalies, or gastrointestinal anomalies such as tracheoesophageal fistula, or necrotizing enterocolitis ,
* receiving xanthine derivatives, H2 blockers, prokinetics, proton pump inhibitors or sedation

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pepsin concentration in tracheal aspirate | 6 hours after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Reem Mahmoud, MD, Principal Investigator — Cairo University Children's Hospital
Locations (1):
- Cairo University Children's Hospital, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Farhath S, He Z, Nakhla T, Saslow J, Soundar S, Camacho J, Stahl G, Shaffer S, Mehta DI, Aghai ZH. Pepsin, a marker of gastric contents, is increased in tracheal aspirates from preterm infants who develop bronchopulmonary dysplasia. Pediatrics. 2008 Feb;121(2):e253-9. doi: 10.1542/peds.2007-0056. PMID 18245400
- [Background] Aly H, Badawy M, El-Kholy A, Nabil R, Mohamed A. Randomized, controlled trial on tracheal colonization of ventilated infants: can gravity prevent ventilator-associated pneumonia? Pediatrics. 2008 Oct;122(4):770-4. doi: 10.1542/peds.2007-1826. PMID 18829800